CLINICAL TRIAL: NCT07088666
Title: Comparison of 0.2% Chlorhexidine and MicroRepair ABX Mouthwash in Patients With Plaque-Induced Gingivitis: A Randomized Controlled Trial
Brief Title: 0.2% Chlorhexidine vs MicroRepair ABX in Gingivitis
Acronym: GEM-CHX02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-CHX0.2vsMICRO
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Gingivitis and Periodontal Diseases; Dental Plaque; Oral Hygiene
Keywords: Chlorhexidine 0.2%; MicroRepair ABX; Gingivitis; Plaque-induced gingivitis; Mouthwash; Oral hygiene; Dental plaque; aMMP-8; Periodontal health; Randomized controlled trial; Non-surgical periodontal therapy
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Dental Plaque | interventions — Chlorhexidine; Mouthwashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MicroRepair ABX Mouthwash (Experimental): Participants assigned to this arm will receive professional dental cleaning at baseline (T0). After this visit, they will use MicroRepair® ABX mouthwash, which contains biomimetic zinc-hydroxyapatite microcrystals enriched with antibacterial agents. The prescribed regimen is 10 mL of mouthwash for 30 seconds, twice daily, for 14 days, after toothbrushing, without rinsing with water for at least 1 hour.
  Follow-up visits will be scheduled at 2 weeks (T1), 1 month (T2), 3 months (T3), and 6 months (T4). At each visit, periodontal parameters and patient-reported outcomes will be recorded. Salivary samples for activated Matrix Metalloproteinase-8 (aMMP-8) analysis will be collected at T0 and T1.
  Interventions: Drug: MicroRepair ABX mouthwash
- 0.2% Chlorhexidine Mouthwash (Active Comparator): Participants assigned to this arm will receive professional dental cleaning at baseline (T0). After this visit, they will use chlorhexidine digluconate 0.2% mouthwash, considered the gold standard for chemical plaque control. The prescribed regimen is 10 mL of mouthwash for 30 seconds, twice daily, for 14 days, after toothbrushing, without rinsing with water for at least 1 hour.
  Follow-up visits will be scheduled at 2 weeks (T1), 1 month (T2), 3 months (T3), and 6 months (T4). At each visit, periodontal parameters and patient-reported outcomes will be recorded. Salivary samples for activated Matrix Metalloproteinase-8 (aMMP-8) analysis will be collected at T0 and T1.
  Interventions: Drug: Chlorhexidine 0.2% mouthwash

INTERVENTIONS:
Drug: MicroRepair ABX mouthwash — At baseline (T0), participants receive clinical assessments, oral hygiene instruction, and begin a 14-day home regimen with MicroRepair® ABX mouthwash, which contains zinc-hydroxyapatite microcrystals and antibacterial agents (cetylpyridinium chloride, magnolol, honokiol). The mouthwash is used twice daily (10 mL for 30 seconds) after toothbrushing, without rinsing, and participants avoid food or drink for 1 hour. All participants use a sodium lauryl sulfate (SLS)-free toothpaste (Biorepair®) throughout the study.
  At 1 month (T1), participants undergo professional supragingival prophylaxis following the Guided Biofilm Therapy (GBT) protocol, which includes plaque disclosure, ultrasonic debridement with an EMS Piezon piezoelectric device, and air-polishing with glycine powder.
  At 3 months (T2) and 6 months (T3), additional GBT sessions and a repeated 14-day mouthwash cycle are performed only if the Full-Mouth Bleeding Score (FMBS) remains greater than 10%.
  Other Names: Hydroxyapatite-based mouthwash
  Arms: MicroRepair ABX Mouthwash
Drug: Chlorhexidine 0.2% mouthwash — At baseline (T0), participants undergo clinical and photographic assessments, receive oral hygiene instruction, and begin a 14-day home regimen with 0.2% chlorhexidine digluconate mouthwash, used twice daily (10 mL for 30 seconds) after toothbrushing. The solution is not rinsed away, and participants avoid food or drink for 1 hour. All participants use a standardized sodium lauryl sulfate (SLS)-free toothpaste (Biorepair®).
  At 1 month (T1), participants receive professional supragingival prophylaxis following the Guided Biofilm Therapy (GBT) protocol, which includes plaque disclosure, piezoelectric ultrasonic scaling with an EMS Piezon device, and air-polishing with glycine powder.
  At 3 months (T2) and 6 months (T3), additional GBT sessions and repetition of the 14-day home regimen are performed only if the Full-Mouth Bleeding Score (FMBS) remains greater than 10%.
  Other Names: Chlorhexidine digluconate 0.2%
  Arms: 0.2% Chlorhexidine Mouthwash

SUMMARY:
Gingivitis is the most common form of reversible gum disease, caused by the accumulation of dental plaque. It leads to inflammation of the gums, bleeding, and discomfort, but it can be managed and reversed with professional dental cleaning and proper oral hygiene.

Chlorhexidine 0.2% mouthwash is considered the "gold standard" in reducing plaque and gingival inflammation. However, its long-term use may cause side effects such as tooth staining, changes in taste, and irritation of the oral tissues. MicroRepair® ABX mouthwash, which contains biomimetic zinc-hydroxyapatite microcrystals with antibacterial components, has shown promising properties in reducing plaque and supporting gum health, with potentially fewer side effects.

This randomized controlled clinical trial will compare the effectiveness of 0.2% chlorhexidine mouthwash and MicroRepair® ABX mouthwash, both used after professional dental cleaning, in patients with plaque-induced gingivitis. Forty participants will be randomly assigned to one of the two treatments for 14 days.

The primary outcome will be the change in gum pocket depth, measured as Probing Pocket Depth (PPD). Secondary outcomes include changes in plaque accumulation, measured as Full-Mouth Plaque Score (FMPS); gum bleeding, measured as Full-Mouth Bleeding Score (FMBS); attachment of the gums to the teeth, measured as Clinical Attachment Level (CAL); gum recession, measured as Recession (REC); tooth staining, measured with the Lobene Stain Index; tooth sensitivity, measured with the Schiff Air Index; taste alterations assessed through a validated questionnaire; and salivary levels of activated Matrix Metalloproteinase-8 (aMMP-8), a biomarker of gum inflammation.

The goal of this study is to determine whether MicroRepair® ABX is as effective as chlorhexidine 0.2% in treating plaque-induced gingivitis, while offering better tolerability and fewer side effects.

DETAILED DESCRIPTION:
Gingivitis is a reversible inflammatory condition of the gums, caused by the accumulation of dental plaque. It is characterized by gum redness, swelling, and bleeding, but it does not involve loss of attachment or bone support. Although it can be effectively managed, untreated gingivitis may progress to periodontitis, which is a more severe and irreversible disease.

Chlorhexidine digluconate 0.2% is widely regarded as the gold standard among antiseptic mouthwashes because of its proven antibacterial and anti-plaque properties. Nevertheless, its long-term use is limited by adverse effects, including tooth and tongue staining, altered taste perception, and mucosal irritation. For this reason, alternative formulations with similar antibacterial potential but fewer side effects are under investigation.

MicroRepair® ABX mouthwash contains biomimetic zinc-hydroxyapatite microcrystals enriched with antibacterial agents. Zinc-hydroxyapatite has shown the ability to reduce plaque accumulation, promote enamel remineralization, and support gum health without cytotoxic effects. Despite encouraging in vitro results and clinical studies in other conditions, there is still a lack of randomized controlled trials directly comparing MicroRepair® ABX with chlorhexidine 0.2% in patients with plaque-induced gingivitis.

This study aims to fill this gap by evaluating whether MicroRepair® ABX is as effective as chlorhexidine 0.2% in reducing gingival inflammation after professional dental cleaning. In addition to standard clinical measures-such as Probing Pocket Depth (PPD), Full-Mouth Plaque Score (FMPS), Full-Mouth Bleeding Score (FMBS), Clinical Attachment Level (CAL), and Recession (REC)-the trial will also assess patient-related outcomes including tooth staining (Lobene Stain Index), dentinal sensitivity (Schiff Air Index), and taste alterations. Furthermore, salivary levels of activated Matrix Metalloproteinase-8 (aMMP-8), a sensitive biomarker of periodontal inflammation, will be analyzed to provide insight into the biological mechanisms of action.

By integrating both clinical and biomolecular outcomes, this study will generate robust evidence on whether MicroRepair® ABX can serve as a safe and effective alternative to chlorhexidine 0.2% in the management of plaque-induced gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 70 years
* Presence of generalized plaque-induced gingivitis (FMBS ≥ 25%, PPD ≤ 3 mm in ≥90% of sites)
* At least 20 natural teeth
* Good general health (ASA I or II)
* Signed written informed consent
* Willingness to comply with study protocol and attend all follow-up visits

Exclusion Criteria:

* Periodontitis (defined as interdental CAL ≥1 mm at ≥2 non-adjacent teeth)
* Systemic diseases affecting periodontal status (e.g., diabetes, immunodeficiencies)
* Antibiotic or anti-inflammatory therapy in the last 3 months
* Professional dental cleaning in the past 3 months
* Pregnancy or breastfeeding
* Known allergy to chlorhexidine or microRepair® components
* Use of orthodontic appliances or removable prostheses
* Smoking more than 10 cigarettes per day
* Participation in other clinical trials in the past 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Change in periodontal probing depth assessed by Probing Pocket Depth (PPD) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  Periodontal probing depth (PPD) is defined as the distance from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, measured in millimeters with a calibrated periodontal probe (Hu-Friedy PCP UNC 15). PPD is assessed at six sites per tooth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual). For each participant, a mean PPD score is calculated at each time point (T0, T1, T2, T3, T4). Possible PPD scores typically range from 1 mm (healthy sulcus) to ≥7 mm (advanced pocket). A higher score indicates more severe gingival inflammation or periodontal attachment loss.
  The primary endpoint is the change in mean PPD from baseline (T0) to 6 months (T4), comparing the two groups: MicroRepair® ABX mouthwash regimen vs chlorhexidine digluconate 0.2% mouthwash regimen. All participants receive supragingival prophylaxis according to the Guided Biofilm Therapy (GBT) protocol.

SECONDARY OUTCOMES:
Change in plaque accumulation assessed by Full Mouth Plaque Score (FMPS) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  The Full-Mouth Plaque Score (FMPS) quantifies the percentage of tooth surfaces with visible dental plaque, assessed after plaque disclosure at four sites per tooth (mesial, buccal, distal, lingual). The score is calculated as the number of plaque-positive sites divided by the total number of sites ×100. Possible scores range from 0% (no plaque) to 100% (plaque on all surfaces). Lower scores indicate better oral hygiene. For each participant, a mean FMPS is calculated at each time point (T0, T1, T2, T3, T4).
Change in gingival inflammation assessed by Full Mouth Bleeding Score (FMBS) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  The Full-Mouth Bleeding Score (FMBS) measures the percentage of bleeding sites after gentle probing at four sites per tooth (mesial, buccal, distal, lingual). FMBS reflects the presence and severity of gingival inflammation. Scores range from 0% (no bleeding) to 100% (bleeding at all sites). A higher FMBS indicates more severe gingival inflammation. For each participant, a mean FMBS is calculated at each time point (T0, T1, T2, T3, T4).
Change in salivary inflammation assessed by activated Matrix Metalloproteinase-8 (aMMP-8) levels | Baseline (T0), 2 weeks (T1)
  Salivary activated Matrix Metalloproteinase-8 (aMMP-8) is a biomarker of periodontal inflammation and collagen breakdown. At baseline (T0) and 2 weeks (T1), unstimulated whole saliva samples are collected using a standardized sterile protocol. Participants refrain from eating, drinking, or brushing their teeth for at least 1 hour before collection. Saliva is collected passively into sterile tubes over 5 minutes, immediately frozen at -20°C, and later analyzed via immunoassay (enzyme-linked immunosorbent assay, ELISA).
  Results are expressed in nanograms per milliliter (ng/mL) and interpreted as: <8 ng/mL = no inflammation; 9-19 ng/mL = mild inflammation; >20 ng/mL = severe inflammation. For each participant, mean aMMP-8 levels will be calculated at T0 and T1.
Change in gingival recession assessed by Recession (REC) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  Gingival Recession (REC) is defined as the distance in millimeters from the cemento-enamel junction (CEJ) to the gingival margin, measured at six sites per tooth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual) using a calibrated periodontal probe (Hu-Friedy PCP UNC 15). Measurements are performed at baseline (T0), after completion of the 14-day mouthwash protocol (T1, 2 weeks), following professional supragingival prophylaxis (T2, 1 month), and during the subsequent follow-up visits (T3, 3 months, and T4, 6 months). Scores range from 0 mm (no recession) to values exceeding 5 mm in cases of severe gingival recession. For each patient, a mean REC score is calculated at every time point (T0-T4) to monitor potential soft tissue loss over the study period. Mean REC values will be compared between the MicroRepair® ABX mouthwash regimen and the chlorhexidine digluconate 0.2% mouthwash regimen.
Change in clinical attachment level assessed by Clinical Attachment Level (CAL) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  Clinical Attachment Level (CAL) is defined as the distance in millimeters from the cemento-enamel junction (CEJ) to the base of the periodontal pocket, recorded at six sites per tooth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual) using a calibrated periodontal probe (Hu-Friedy PCP UNC 15). Measurements are performed at baseline (T0), after completion of the 14-day mouthwash regimen (T1, 2 weeks), following professional supragingival prophylaxis (T2, 1 month), and at subsequent follow-up visits (T3, 3 months, and T4, 6 months). CAL values typically range from 0 mm (healthy periodontium) to ≥7 mm (advanced attachment loss). For each patient, a mean CAL score is calculated at every time point (T0-T4). Mean CAL values will be compared between the MicroRepair® ABX mouthwash regimen and the chlorhexidine digluconate 0.2% mouthwash regimen to assess differences in periodontal tissue attachment loss.
Change in extrinsic staining assessed by Lobene Stain Index Modified | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  The Modified Lobene Stain Index is used to evaluate extrinsic dental staining on vestibular and lingual/palatal tooth surfaces by assessing both stain intensity and extent. Intensity is scored as 0 = no stain, 1 = light stain, 2 = moderate stain, and 3 = heavy stain. Extent is scored as 0 = no stain, 1 = stain covering up to one-third of the surface, 2 = stain covering between one-third and two-thirds of the surface, and 3 = stain covering more than two-thirds of the surface. The final score for each surface is obtained by multiplying intensity by extent, with higher scores indicating more pronounced staining. Assessments are conducted at baseline (T0), after completion of the 14-day mouthwash regimen (T1, 2 weeks), following professional supragingival prophylaxis (T2, 1 month), and during subsequent follow-up visits (T3, 3 months, and T4, 6 months). The index is used to compare the staining potential of the MicroRepair® ABX mouthwash regimen versus the chlorhexidine digluconate 0.2%
Change in dentin hypersensitivity assessed by Schiff Air Index | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  The Schiff Air Index is employed to assess dentin hypersensitivity in response to a standardized air stimulus directed onto the vestibular surface of each tooth. Responses are scored as 0 = no response, 1 = response without request to discontinue the stimulus, 2 = response with a request to discontinue the stimulus, and 3 = painful response with immediate withdrawal or visible discomfort. For each patient, a mean Schiff score is calculated at every evaluation. Measurements are performed at baseline (T0), after completion of the 14-day mouthwash regimen (T1, 2 weeks), following professional supragingival prophylaxis (T2, 1 month), and during the follow-up visits (T3, 3 months, and T4, 6 months). Scores will be compared between the MicroRepair® ABX mouthwash regimen and the chlorhexidine digluconate 0.2% regimen to determine the impact of treatments on dentin hypersensitivity over time.
Change in taste perception assessed by a validated taste alteration questionnaire | 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  Taste perception will be assessed using a validated patient-reported questionnaire designed to capture the presence and severity of taste alterations, including bitter, metallic, or unpleasant sensations. Each item is scored on a 5-point Likert scale, where 0 = no alteration, 1 = mild alteration, 2 = moderate alteration, 3 = severe alteration, and 4 = very severe alteration. For each patient, a total score is calculated, with higher values indicating more pronounced dysgeusia. Evaluations are performed at baseline (T0), after completion of the 14-day mouthwash regimen (T1, 2 weeks), following the first professional supragingival prophylaxis (T2, 1 month), and during follow-up visits (T3, 3 months, and T4, 6 months). Mean scores will be compared between the MicroRepair® ABX mouthwash regimen and the chlorhexidine 0.2% regimen to assess and compare the tolerability of the interventions over time.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.